CLINICAL TRIAL: NCT01844089
Title: The Use of the Bakri Postpartum Balloon in the Management of Postpartum Hemorrhage Refractory to Conservative Measures: A Multi-Site Longitudinal Study An Initiative Under the East African Women's Health Network (EAWoHNet)
Brief Title: The Use of the Bakri Postpartum Balloon in the Management of Postpartum Hemorrhage Refractory to Conservative Measures
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00029944
Record Dates: First submitted 2013-04-29; First posted 2013-05-01 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum hemorrhage; Bakri Postpartum Balloon
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The broad objective of the study is to determine if the Bakri Postpartum Balloon is effective in preventing morbidity and mortality from postpartum hemorrhage (PPH) as part of a standardized management algorithm.

Specific Objectives

* To estimate the rate of morbidity (including operative intervention and peripartum hysterectomy) and mortality secondary to PPH in 4 academic centers after introduction of a standardized protocol for management of PPH, but prior to the inclusion of the Bakri Postpartum Balloon as part of the protocol.
* To estimate the rate of morbidity (including operative intervention and peripartum hysterectomy) and mortality secondary to PPH in 4 academic centers after introduction of a standardized protocol for management of PPH, after the inclusion of the Bakri Postpartum Balloon as part of the protocol.
* To compare morbidity
* To generate preliminary data for (a) a larger confirmatory study of the use of the Bakri Postpartum Balloon in centers with surgical and blood transfusion services, and (b) design of a pilot study of the use of the Bakri device of temporary control of PPH in settings outside of surgical centers (such as by trained midwives or emergency transport personnel).

DETAILED DESCRIPTION:
Phase I: Development and training of staff in standardized algorithm for management of PPH using available local resources (not including Bakri balloon).

Phase II: Data collection after introduction of the standardized algorithm.

Phase III: Revision of protocol to include the Bakri Postpartum Device

Phase IV: Data collection after introduction of the Bakri device

Bakri Postpartum Balloon 510K Premarket Notification/Cook OBGYN #K062438

ELIGIBILITY:
Inclusion Criteria:

* Any woman who recently delivered by either vaginal or cesarean delivery who experiences postpartum hemorrhage, defined as
* Clinically estimated blood loss of greater than 500 ml for a vaginal delivery, or
* Clinically estimated blood loss of greater than 1000 ml for a cesarean delivery, or
* Hemodynamic changes that, in the opinion of the care team, require interventions beyond routine postpartum or postdelivery care (such as intravenous fluids or the use of more than one uterotonic agent).

Exclusion Criteria:

* Minors (less than 18 years of age)
* Arterial bleeding requiring surgical exploration or angiographic embolization
* Cases requiring immediate lifesaving hysterectomy
* Ongoing intrauterine pregnancy
* Cervical cancer
* Purulent infections of the vagina, cervix or uterus
* Untreated uterine anomaly
* Disseminated intravascular coagulation
* A surgical site which would prohibit the device from effectively controlling bleeding
* Patients who are referred for obstructed labor
* Patients with signs, symptoms or other evidence of ruptured uterus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any woman who recently delivered by either vaginal or cesarean delivery who experiences postpartum hemorrhage.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Composite clinical outcome | 24 hours
  The primary outcome of the study is a composite clinical outcome consisting of:
  * Blood transfusion
  * Renal failure (creatinine >1.5 mg/dL or increased >1.0 mg/dL above baseline, oliguria <120 ml output in 4 hour intervals)
  * Respiratory impairment (impairment of respiratory function requiring ventilation, oxygen supplementation, or decreased physical activity compared to pre-pregnancy levels)
  * Central nervous system impairment (seizures, loss of consciousness, or cognitive/motor loss)
  * Heart failure (NYHA class III or IV)
  * Disseminated intravascular coagulation (DIC) based on clinical and laboratory assessment if available.
  * Abdominal surgery to control hemorrhage in non-cesarean patients
  * Emergency hysterectomy. Outcomes and definitions are similar to those used in other studies of PPH management in Africa.

SECONDARY OUTCOMES:
Unit of estimated blood loss | 24 hours
  Mean and median estimated blood loss

OTHER OUTCOMES:
Number of women with febrile morbidity | 24 hours
  febrile morbidity and individual rates of the components of the composite primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Haywood Brown, MD, Principal Investigator — DUHS
Locations (2):
- Kenya (2):
  - MOI Teaching and Referral Hospital, Eldoret
  - Great Lakes University, Kisumu